CLINICAL TRIAL: NCT03964506
Title: A Pilot Study to Determine the Safety and Efficacy of Incorporating Hyperbaric Oxygen Therapy Into RIC Fludarabine and Melphalan and Allogeneic Hematopoietic Stem/Progenitor Transplantation
Brief Title: Hyperbaric Oxygen Therapy and Allogeneic Peripheral Blood Stem Cell (PBSC) Transplant
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Omar Aljitawi (Other)
Responsible Party: Sponsor-Investigator, Omar Aljitawi, Associate Professor of Hematology/Oncology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBMT-19163
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Atypical Chronic Myeloid Leukemia; Chronic Monocytic Leukemia; Myelofibrosis; Myelodysplastic/Myeloproliferative Neoplasm
Keywords: Allogeneic transplant; Hyperbaric Oxygen
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myeloid; Primary Myelofibrosis; Myelodysplastic-Myeloproliferative Diseases | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1- AML or MDS (Experimental): Patients with will receive HBO therapy one time on day 0 of the transplant. The treatment consists of exposure to hyperbaric oxygen at 2.5 atmospheric absolutes (ATA) for a total of 90 minutes after compression to 2.5 atmosphere absolutes (ATA) in a monoplace hyperbaric chamber (Model 3200/3200R, Sechrist Industries, Inc., USA), breathing 100% oxygen. The subjects will be in the chamber for a total of 120 minutes as approximately 10-15 minutes were spent during the compression and decompression phases and subjects had 10 minute room air breaks every 30 minutes of hyperbaric oxygen treatment.
  Interventions: Drug: Hyperbaric oxygen
- Cohort 2- CMML, aCML, CML, CNL, MDS/MPN (Experimental): Patients with will receive HBO therapy one time on day 0 of the transplant. The treatment consists of exposure to hyperbaric oxygen at 2.5 atmospheric absolutes (ATA) for a total of 90 minutes after compression to 2.5 atmosphere absolutes (ATA) in a monoplace hyperbaric chamber (Model 3200/3200R, Sechrist Industries, Inc., USA), breathing 100% oxygen. The subjects will be in the chamber for a total of 120 minutes as approximately 10-15 minutes were spent during the compression and decompression phases and subjects had 10 minute room air breaks every 30 minutes of hyperbaric oxygen treatment.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — Reduced intensity conditioning Fludarabine and Melphalan with Hyperbaric Oxygen and Allogeneic Hematopoietic Stem Cell Transplant
  Other Names: HBO

SUMMARY:
The purpose of this study is to determine if hyperbaric oxygen therapy is safe in the setting of stem cell transplantation. This study will also determine if hyperbaric oxygen therapy improves engraftment, graft versus host disease, neutrophil count, and incidence and severity of mucositis (inflammation of the mouth or gut) and infection. This study has two cohorts. The first cohort is subjects with acute myeloid leukemia (AML) or Myelodysplastic Syndrome (MDS). The second cohort is subjects with chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), chronic monocytic leukemia, chronic neutrophilic leukemia (CNL), myelofibrosis, and myelodysplastic/myeloproliferative (MDS/MPN) overlap syndrome. The first cohort has completed the recruitment so only the second cohort will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent
* Men or women, age ≥ 18 years of age, with upper limit of 75 years old.
* Subjects with acute myeloid leukemia (AML) or Myelodysplastic Syndrome (MDS) for cohort 1.
* Subjects with chronic myelomonocytic leukemia (CMML), atypical chronic myeloid leukemia (aCML), CML, chronic neutrophilic leukemia (CNL), myelofibrosis, and myelodysplastic/myeloproliferative (MDS/MPN) overlap syndrome for cohort 2.
* Karnofsky performance status (KPS) of ≥ 70%
* Patients should have New York Heart Association (NYHA) Functional Classification, Class I (ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain) or Class II (ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain).
* Adequate hepatic, renal, cardiac and pulmonary function to be eligible for transplant. Minimum criteria include: Hepatic: ALT, AST < 4x IULN and serum total bilirubin ≤ 2.0 mg/dL; Renal: serum creatinine: ≤ 2.0 mg/dL; Left ventricular ejection fraction ≥ 45% measured by 2D-ECHO or MUGA scan; EKG with no clinically significant arrhythmia; FEV1, FVC and DLCO ≥ 50% of predicted value (corrected to serum hemoglobin)
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days following completion of therapy. Should a woman or partner become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician and the investigator immediately.
* A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Women of child-bearing potential should have a negative urine or serum pregnancy test within 4 weeks of starting preparative regimen

Exclusion Criteria:

* Pregnant or breastfeeding
* Severe chronic obstructive pulmonary disease requiring oxygen supplementation
* History of spontaneous pneumothorax, prior chest surgery requiring thoracotomy or direct chest irradiation to the lungs
* Evidence of pneumothorax or significant pulmonary fibrosis on chest imaging within 60 days of transplant.
* Active malignancy excluding AML, MDS, CMML, aCML CML, CNL, MF and MDS/MPN overlap syndrome.
* Active ear/sinus infection. Patients with chronic sinusitis or sinus headaches are excluded unless cleared by ear, nose, and throat specialist.
* Recent sinus surgery (within the last 5 years).
* Ear surgery excluding myringotomy or ear tubes
* Subjects must agree to refrain from active tobacco or e-cigarette use 72 hours prior to transplant until complete transplant recovery. Nicotine replacement therapy is allowed.
* Claustrophobia
* History of recurrent seizures within 5 years of study enrollment.
* Uncontrolled asthma
* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 months) invasive fungal infection without interdisciplinary (ID) consult and approval
* Patients who had intrathecal chemotherapy within 2 weeks of starting preparative regimen or cranial irradiation within 4 weeks of starting preparative regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Immediate safety of hyperbaric oxygen therapy prior to allogeneic stem cell transplantation in Cohort 1 | 24 hours
  Treatment-limiting toxicities will be assessed 24-hours post-hyperbaric oxygen therapy.
Immediate safety of hyperbaric oxygen therapy prior to allogeneic stem cell transplantation in cohort 2 | 24 hours
  Treatment-limiting toxicities will be assessed 24-hours post-hyperbaric oxygen therapy.
Long term safety of hyperbaric oxygen therapy prior to allogeneic stem cell transplant in Cohort 1 | 100 days
  Possible long-term effects of hyperbaric oxygen therapy treatment prior to allogeneic peripheral blood stem cell transplant will be assessed at day +100 post-transplant
Long term safety of hyperbaric oxygen therapy prior to allogeneic stem cell transplant in Cohort 2 | 100 days
  Possible long-term effects of hyperbaric oxygen therapy treatment prior to allogeneic peripheral blood stem cell transplant will be assessed at day +100 post-transplant

SECONDARY OUTCOMES:
Time to neutrophil recovery in Cohort 1 | 100 days
  based on the patient having achieved three consecutive days of Absolute Neutrophile Count (ANC) ≥ 500/microliter
Time to neutrophil recovery in Cohort 2 | 100 days
  based on the patient having achieved three consecutive days of Absolute Neutrophile Count (ANC) ≥ 500/microliter
Time to complete donor chimerism in Cohort 1 | 100 days
  Bone marrow chimerism will be checked on day +30 and day +100 Bone Marrow (BM) samples according to our standard of care
Time to complete donor chimerism in Cohort 2 | 100 days
  Bone marrow chimerism will be checked on day +30 and day +100 Bone Marrow (BM) samples according to our standard of care
Incidence of mucositis in Cohort 1 | 100 days
Incidence of graft versus host disease in Cohort 1 | 100 days
Incidence of infection in Cohort 1 | 100 days
Incidence of mucositis in Cohort 2 | 100 days
Incidence of infection in Cohort 2 | 100 days
Incidence of graft versus host disease in Cohort 2 | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Omar S Aljitawi, MBBS, Principal Investigator — University of Rochester
Locations (1):
- Wilmot Cancer Institute, University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial will be shared after deidentification, including dictionaries.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data for any type of analyses.